CLINICAL TRIAL: NCT06981468
Title: H2O - Hydration to be Optimized With a Low-sodium Beverage
Brief Title: Hydration To be Optimized (H2O) With a Low-sodium Beverage
Acronym: H2O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2309NR
Record Dates: First submitted 2025-04-23; First posted 2025-05-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hydration Status
Keywords: Hydration; Low-sodium beverage; H20
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional Product 1 (Active Comparator): Glycerol (Dose 1) and Whey Protein
  Interventions: Dietary Supplement: Low Sodium Beverage 1
- Interventional Product 2 (Active Comparator): Glycerol (Dose 2) and Whey Protein
  Interventions: Dietary Supplement: Low Sodium Beverage 2
- Comparator (Placebo Comparator): Water
  Interventions: Other: Control (placebo) group

INTERVENTIONS:
Dietary Supplement: Low Sodium Beverage 1 — The first interventional product for this study is a low-sodium beverage containing Dose 1 of glycerol, whey protein, and water. It will come in a ready to drink format for the participants.
  Arms: Interventional Product 1
Dietary Supplement: Low Sodium Beverage 2 — The second interventional product for this study is a low-sodium beverage containing dose 2 of glycerol, whey protein, and water. It will come in a ready to drink format for the participants.
  Arms: Interventional Product 2
Other: Control (placebo) group — Water
  Arms: Comparator

SUMMARY:
In this study, the investigators want to assess the effects of a new beverage containing whey protein and glycerol (two different dosages) on hydration status in healthy adults when compared to the control (water).

This is a single-center, double-blinded, 3 arm cross-over randomized controlled study looking to enroll 45 healthy adult participants. The study will be performed at the Clinical Innovation Lab (CIL), Nestlé Research, Lausanne. Participants will be screened and randomly assigned to 1 of 6 sequences of consumption. Enrolled participants will have three visit days. They will consume one of the test products, or control at each visit and complete the study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male adults aged 18-50 years.
2. Body mass index (BMI) between 18.5 to 25 kg/m² (inclusive).
3. Healthy as determined based on self-reported medical history.
4. Able to understand and to sign a written informed consent prior to study enrolment.
5. Willing and able to comply with the requirements for participation in this study.

Exclusion Criteria:

1. Any past or on-going diagnosed medical/surgical condition (e.g. malignancy, renal condition, liver condition, uncontrolled diabetes mellitus, cardiovascular disease, hypertension, migraine and headache disorders) and/ or psychiatric condition (e.g. depression, psychotic disorders, chronic insomnia, eating disorder), which in the opinion of the site physician/investigator may risk participant's well-being/safety, impede participant compliance with study procedures or ability to complete the study and/or could confound the primary objectives of the study.
2. Current intake of medication/s that impact hydration status (e.g. anti-hypertensive medications, anti-diabetic medications, anti-psychotics, anti-depressants, diuretics, laxatives, antidiuretic hormone (ADH) antagonists, oral corticosteroids, glucocorticoids, anti-cholinergic medications, or cyclosporine A).
3. Currently on a high-protein (1.5g/kg/BW/day) or ketogenic diet (based on self-report).
4. Known/suspected food allergy or intolerance to any food (based on self-report).
5. Female participants who are pregnant, lactating and/or breastfeeding (self-report or if in doubt, via urine pregnancy test).
6. Any self-reported chronic alcohol or drug abuse within the past year; specifically, an average alcohol intake > 2 standard drinks per day over a week for males, and > 1 standard drink per day over a week for females. One standard drink contains 10-12 g of ethanol, i.e., 0.3 dl of strong alcohols, 1dl of wine, 3 dl of beer.
7. Currently participating in another interventional study.
8. Family or hierarchical relationships with the research team members.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Fluid Retention (%) - fluid intake vs. urine output measurement | From Baseline (Timepoint 0 minutes) to 2hrs after baseline (Timepoint 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  Difference in fluid retention 2 hours after intake of the study product in comparison with the control by measuring urine output in comparison to fluid intake.

SECONDARY OUTCOMES:
Fluid Retention (%) 1hr measure - fluid intake vs. urine output measurement | From Baseline (Timepoint 0 minutes) to 1hr after baseline (Timepoint 60 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  Difference in fluid retention 1 hour after intake of the study product in comparison with the control by measuring urine output in comparison to fluid intake.
Fluid Retention (%) between interventional products - fluid intake vs. urine output measurement | From Baseline(Timepoint 0 minutes), to 1hr after baseline (Timepoint 60 minutes), and to 2hrs after baseline (Timepoint 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  Difference in fluid retention at 1hour and 2hours after intake of the study product, comparing both study products containing the different doses of glycerol.
Net Fluid Balance - fluid intake vs. urine output measurement, weighted on the scale | From Baseline (Timepoint 0 minutes) to 1hr after baseline(Timepoint 60 minutes), and at 2hrs after baseline (Timepoint 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  Net fluid balance at 1 hour and 2 hours after intake of study product, comparing the study products with the control, and between both study products containing different doses of glycerol.
Urine weight - weighted on the scale | From Baseline (Timepoint 0 minutes) to 1hr after baseline (Timepoint 60 minutes), and at 2hrs after baseline (Timepoint 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  Urine weight at 1 hour after intake and cumulative urine weight after 2 hours of intake of the study product, comparing the study products with the control, and between both study products containing different doses of glycerol.
Cumulative Urine Weight - weighted on the scale | From Baseline (Timepoint 0 minutes) and at 2 hrs after baseline (Timepoint 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  The cumulative urine weight 2 hours after intake of the study products relative to the cumulative urine weight 2 hours after intake of the control (Beverage Hydration Index [BHI]), comparing both study products containing different doses of glycerol.
Urine Specific Gravity (USG) - measured in duplicate with a Digital Hand-Held Pen-Pro Refractometer (Atago 3730) | From Baseline (Timepoint 0 minutes) to 1hr after baseline (Timepoint 60 minutes), and at 2hrs after baseline (Timepoint 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  USG 1 and 2 hours after intake of the study product, comparing the study products with the control, and between both study products containing different doses of glycerol.
Change in USG from baseline to 1 and 2 hours - measured in duplicate with a Digital Hand-Held Pen-Pro Refractometer (Atago 3730) | From Baseline (Timepoint 0 minutes) to 1hr after baseline (Timepoint 60 minutes), and at 2hrs after baseline (Timepoint 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  Change in USG from baseline to 1 and 2 hours after intake (delta0-60min, delta0-120min) after intake of the study product, comparing the study products with the control, and between both study products containing different doses of glycerol.
Change in calculated serum osmolality - by Blood Microsampling with Tasso Device | From Baseline (Timepoint 0 minutes), to 30min after baseline (Timepoint 30 minutes), to 1hr after baseline (Timepoint 60 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7)
  Change in calculated serum osmolality during 30-minute and 1 hour after intake of the study products, comparing the study products with the control, and between both study products containing different doses of glycerol.
Hydration Questionnaire Part 1 - Visual Analogue Scale (VAS) Questionnaire (From 0-10cm, 0 indicating "not at all" and 10 indicating "extremely") | From Baseline (Timepoint 0 minutes), to 30min after baseline (Timepoint 30 minutes), to 1hr after baseline (Timepoint 60 minutes), and 2hrs after baseline (Timepoints 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7).
  Hydration Questionnaire Part 1 Visual Analogue Scale (VAS) scores at 30 minutes, 1 hour, and 2 hours after intake of the study product, comparing the study products with the control, and between both study products containing different doses of glycerol.
Hydration Questionnaire Part 2 - Visual Analogue Scale (VAS) Questionnaire (Scale 0-10 cm, 0 indicating the worst score and 10 indicating the best score) | 5 minutes after Baseline (Timepoint 5 minutes), at 2 hrs after baseline (Timepoint 120 minutes), at Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7).
  Hydration Questionnaire Part 2 ratings, comparing the study products with the control, and between both study products containing different doses of glycerol.
Safety and Tolerability - Beverage Tolerability Questionnaire (Scale of 1-4, 1 indicating no symptoms and 4 indicating severe symptoms) | Prior to Baseline (Upon arrival on-site, before product intake), and at 2 hours after baseline (Timepoint 120 minutes), for Visit 1 (day 3), Visit 2 (day 5), and Visit 3 (day 7).
  Comparison of Beverage Tolerability Questionnaire (BTQ): individual score and composite score between control and study products, and between both study products containing different doses of glycerol.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Schneider, Principal Investigator — Nestlé Research
Locations (1):
- Clinical Innovation Lab, Nestlé Research, Lausanne, Switzerland